CLINICAL TRIAL: NCT04675814
Title: Prospective Evaluation of the Impact on Patients' Quality of Life of a 12-Week Adapted Physical Activity Program (APA) at Institut de Cancerologie de l'Ouest (ICO)
Brief Title: Prospective Evaluation of the Impact on Patients' Quality of Life of a 12-Week Adapted Physical Activity Program (APA)
Acronym: APA
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2020-05
Record Dates: First submitted 2020-12-01; First posted 2020-12-19 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2021-05

CONDITIONS: Sports Physical Therapy
Keywords: Adapted Physical Activity program (APA); kinesiophobia; Fatigue; Quality of life
MeSH Terms: conditions — Kinesiophobia; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adapted Physical Activity (APA) — Adults participating in the APA program at ICO during the first semester of 2020, regardless of cancer type and ongoing treatment (chemotherapy, radiotherapy, hormone therapy, immunotherapy). The APA program duration is : 12 weeks

SUMMARY:
The objective of this study is to evaluate the effects of regular physical practice on fatigue, quality of life and kinesiophobia in patients treated at the ICO in Angers, regardless of the type of cancer and the type of treatment.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effects of regular physical practice on fatigue, quality of life and kinesiophobia in patients treated at the ICO in Angers, regardless of the type of cancer and the type of treatment.

A 12-week Adapted Physical Activity program (APA) is proposed to patients included in the study with an assessment of fatigue, quality of life, level of physical activity and kinesiophobia (fear of movement) at the beginning of the study.

A second assessment of fatigue and quality of life will be done during the 6-week management.

At the end of the program, a final evaluation of fatigue, quality of life and kinesiophobia will be done.

ELIGIBILITY:
Inclusion Criteria:

1. Oncological care at the ICO
2. All types of cancer
3. Regardless of the type of treatment (chemotherapy, radiotherapy, hormone therapy, immunotherapy)
4. Age > 18 years old
5. Follow the APA program at the ICO
6. Subject informed of the study

Exclusion Criteria:

1. Contraindication to the practice of sport
2. APA Program outside the ICO
3. Subject opposing the use of his data
4. Minor or adult patient under guardianship or curatorship
5. Pregnant woman
6. Altered general condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in the ICO's APA program during the enrolment period regardless of the type of cancer and the type of treatment in progress (chemotherapy, radiotherapy, hormone therapy, immunotherapy) who accept to participate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie ABADIE-LACOURTOISIE, MD, Study Chair — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancérologie de L'Ouest, Angers, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date first signed consent: 14 SEP 2020 Date of first patient inclusion: 14 SEP 2020 End of trial date (last visit of last patient): 14 MAR 2021
Pre-assignment Details: All screened patients have been included
Groups:
- Adapted Physical Activity (APA): Adults participating in the APA program at ICO during the first semester of 2020, regardless of cancer type and ongoing treatment (chemotherapy, radiotherapy, hormone therapy, immunotherapy).
Period: Overall Study
Arm/Group | Adapted Physical Activity (APA)
Started | 37
Completed | 33
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Performance status alteration not related to study procedure | 1

BASELINE CHARACTERISTICS:
Population: Cancer patients
Arm/Group | Adapted Physical Activity (APA)
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 37

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life of Patients Participating in the 12-week Adapted Physical Activity Program.
Description: Describe the evolution of the quality of life of patients being treated for their cancer pathology at the ICO site in Angers, and participating in the 12-week adapted physical activity program at ICO.
  Quality of life is measured with the FACIT-F Fatigue and Quality of Life Questionnaire. The questionnaire is structured into five sections, each containing between 6 and 13 items. In total, it includes 40 items, each scored from 0 to 4:
  0 - Not at all
  1. - A little
  2. - Moderately
  3. - Quite a bit
  4. - Very much By adding up the answers, the score range obtained is: 0 to 160. The higher the score, the less tired the patient is.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adapted Physical Activity (APA)
Number analyzed (Participants) | 33
score on a scale | 117.6 (23.5)

2. Secondary Outcome: Describe Attendance at the APA Program.
Description: The number of sessions is planned by the APA coach at the beginning of the APA program. The number of performed sessions is measured.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Number of APA sessions
Arm/Group | Adapted Physical Activity (APA)
Number analyzed (Participants) | 37
Number of APA sessions | 14.2 (6.3)

3. Secondary Outcome: Measure the Evolution of Kinesiophobia (Fear of Movement).
Description: Kinesiophobia is measured with the TAMPA Scale for Kinesiophobia (TSK-CF). This scale assesses the kinesiophobia index presented by the patient at the time of the assessment. The higher the score, the greater the level of kinesiophobia. Total score range: 17 to 68. Higher scores indicate greater fear of movement.
  A score ≥ 40 is considered significant kinesiophobia.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adapted Physical Activity (APA)
Number analyzed (Participants) | 33
score on a scale | 34.45 (6.02)

4. Secondary Outcome: Measure Physical Activity at the Initiation of the APA Program.
Description: The level of physical activity (PA) is assessed using the GPAQ questionnaire. The questionnaire consists of 16 items. Physical activity is expressed in MET-minutes per week (Metabolic Equivalent of Task), calculated from reported activity.
  Based on the score, three profiles are defined:
  High
  * ≥3 days vigorous activity (≥1500 MET-min/week) OR
  * ≥7 days walking/moderate/vigorous PA (≥3000 MET-min/week) Moderate
  * ≥20 min vigorous PA / day, ≥3 days/week OR
  * ≥30 min moderate PA/walking / day, ≥5 days/week OR
  * ≥5 days mixed activity (≥600 MET-min/week) Low
  * Does not meet above criteria
Time Frame: Week 0
Measure: Count of Participants; unit: Participants
Arm/Group | Adapted Physical Activity (APA)
Number analyzed (Participants) | 37
Participants
  High activity level | 1
  Moderate activity level | 19
  Low activity level | 17

ADVERSE EVENTS:
Description: This is a non-interventional (observational) category 3 study. No adverse events (AEs), serious adverse events (SAEs) or all-cause mortality were collected.
  "0" Total Number of Participants at Risk in adverse events, serious adverse events and all-cause mortality sections means that these events were not collected or assessed as part of the study.
Arm/Group | Adapted Physical Activity (APA)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT04675814/Prot_SAP_000.pdf